CLINICAL TRIAL: NCT03600506
Title: Dexmedetomidine as an Adjuvant to General Anesthesia in Patients Undergoing Elective Abdominal Hysterectomy
Brief Title: Dexmedetomidine Adjuvant to General Anesthesia of Abdominal Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed A Elsadany, MD, Principal Investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 3400
Record Dates: First submitted 2018-06-26; First posted 2018-07-26 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Effect of Drugs
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Intervention drug of the study
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Normal Saline (Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive infusion of study drug intravenously 10 minutes before induction of anesthesia as 1 mcg/kg over 10 min followed by 0.4 mcg/kg/hr till the start of wound closure.
  Other Names: Selective α2-agonist sympatholytic drug
  Arms: Dexmedetomidine
Drug: Placebo — Fifty ml of Placebo (normal saline) will be prepared and given intravenously by a syringe pump over 10 minutes initially and then over 1 hour till the start of wound closure.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
To assess the effect of perioperative Dexmedetomidine infusion on Interleukin 6 and cortisol level in patients undergoing general anesthesia for total abdominal hysterectomy

DETAILED DESCRIPTION:
Following the departmental research committee approval and informed patient's consent, 52 patients, undergoing abdominal hysterectomy in Suez Canal University Hospital, will be randomly assigned to one of the two groups (Dexmedetomidine and Placebo) using a table of random numbers.

Patients will be fasting for 6 - 8 hours. All patients will receive oral Midazolam (7.5 mg), and oral Ranitidine (150mg) administered 90 min before arrival in the operating room with a sip of water.

All patients will receive before induction, normal saline 10 ml/kg body weight over 10-15 minutes. Subsequently, intravenous fluid administration will be done according to the need of each patient.

All operations will start between 08:30 am and 09:30 am, to minimize variations in cortisol level.

All patients will receive the Drug of study 10 minutes before induction of anesthesia till the start of wound closure in the form of:

Group (D): Dexmedetomidine 1 mcg/kg over 10 min followed by 0.4 mcg/kg/hr. Group (C): Normal saline prepared in a syringe with the same volume as Dexmedetomidine to assure blinding.

Doses will be calculated, diluted in 50 ml of normal saline and given intravenously by a syringe pump over 10 minutes initially and then over 1 hour till the start of wound closure.

All drugs of the study will be prepared by an independent anesthesiologist who will not share in the study and then selected and given by another one blinded for the content of each syringe.

Airway devices, anesthesia machine, ventilator, flowmeters and monitors will be checked promptly.

Another wide-bore I.V cannula will be inserted in case of blood transfusion.

Monitoring equipment's (Datex-Ohmeda™) will be attached to the patient including 3-leads ECG, non-invasive arterial blood pressure, pulse oximeter and capnograph after tracheal intubation.

The depth of anesthesia will be monitored with Entropy device. The Entropy electrodes will be placed on the forehead and on the lateral angle of orbit and connected to (Datex-Ohmeda™). The target Entropy range will be 40-60 for surgical anesthesia.

Induction of anesthesia will be performed by Propofol 2 mg/kg followed by cis-atracurium 0.15 mg/kg and fentanyl 1 mcg/kg given intravenously after pre-oxygenation with 100% oxygen for at least 3 minutes.

Patients will be manually ventilated with 100% oxygen till intubation after 2 min and with Entropy value of 60 to 40 by Macintosh laryngoscope and appropriate size endotracheal tube.

Maintenance of anesthesia will be carried out by isoflurane varying its end tidal concentration to keep Entropy in the range of 55 to 40 with Air:Oxygen mixture 0.3 fraction of oxygen and flow rate of 2 liters/minute in completely closed circuit.

Cis-atracurium 0.03 mg/kg guided by neuromuscular monitor Train Of Four (TOF) will be used for muscle relaxation.

Hemodynamics (mean arterial blood pressure and heart rate) will be maintained within 25 % of baseline measures.

Any increase of MAP or HR more than 25% of baseline measures on two consecutive readings within 2-3 min will be managed by I.V bolus of Fentanyl 0.5 mcg/kg and any decrease of MAP or HR less than 25 % on two consecutive readings within 2-3 min will be managed by I.V bolus of ephedrine 5 mg or atropine 0.5 mg respectively.

The infusion of study medication will be discontinued if the hypotension persisted > 5 minutes after these interventions upon return of the MAP or HR to within 25% of the baseline value, the study medication infusion will be resumed at 50% of the initial infusion rate and then gradually increased to the initial infusion rate.

The infusion of study medication will be discontinued at the start of wound closure. Upon completion of wound closure, isoflurane will be discontinued and the flow rate will be increased to 5 L/min of 100% Oxygen and residual neuromuscular block will be reversed with neostigmine, 0.05 mg/kg IV, and atropine 0.25 mg/kg IV. The trachea will be extubated when the patient is fully awake. Transfer to the recovery room will be done when the patient scored 7 and above using the modified Aldrete scoring system.

On emergence from anesthesia and immediately in post anesthesia care unit, analgesic regimen, consisting of intravenous patient-controlled morphine analgesia (bolus 1mg, 10-min lockout, maximum dose 5 mg / h), will be used in all groups.

The whole technique and anesthetic procedures will be performed by the same anesthesiologist to avoid as much as possible the inter-individual skill variations.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status Grade I = (normal healthy patients)
* American Society of Anesthesiology physical status Grade II = (patients with mild systemic disease and no functional limitations)
* Patients scheduled for abdominal hysterectomy.

Exclusion Criteria:

* Pre-operative regular medication with opioids and benzodiazepines, alcohol abuse, known sleep disturbance, known endocrine disease.
* Known allergy to Dexmedetomidine.
* Heart block greater than first degree.
* Medication known to affect the sympathetic response or hormonal secretion.
* Smokers

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Interleukin 6 (IL6) | At starting drug infusion (10 minutes before induction of anesthesia) and then 2 hours after induction of anesthesia and 6 hours postoperatively
  Measurement of Serum Serum Interleukin 6 in picogram / milliliter

SECONDARY OUTCOMES:
Change in Serum Cortisol | At starting drug infusion (10 minutes before induction of anesthesia) and then 2 hours after induction of anesthesia and 6 hours postoperatively
  Measurement of Serum Cortisol in microgram/ deciliter
Change in Mean arterial blood pressure | Mean Arterial Blood Pressure before starting infusion of the study drug, immediately before induction and 1, 2, 3 and 5 min after intubation, then immediately before extubation, 1, 2, 3 and 5 min after extubation
  Changes in Mean Arterial Blood Pressure (MABP) in mmHg (not systolic or diastolic) with intubation, extubation and throughout surgery
Change in Heart Rate (HR) | HR before starting infusion of the study drug, immediately before induction and 1, 2, 3 and 5 min after intubation, then immediately before extubation, 1, 2, 3 and 5 min after extubation
  Changes in Heart Rate (HR) with intubation, extubation and throughout surgery
Morphine Consumption in patient controlled analgesia (PCA) | Twenty four hours after attachment of patient controlled analgesia in postoperative care unit
  Morphine Consumption in PCA in first 24 hours postoperatively in mg
Fentanyl consumption in microgram using questionnaire | During intraoperative time
  Total intraoperative Fentanyl consumption in microgram
Isoflurane in milliliter using the Ventilator reading | During intraoperative time
  Total intraoperative Isoflurane consumption in ml
Ephedrine in milligram using quessionnaire | During intraoperative time
  Total amount of ephedrine in mg given because of hypotension and number of times of discontinuation of study medication.
Atropine in milligram using quessionnaire | During intraoperative time
  Total amount of Atropine in mg given because of bradycardia and number of times of discontinuation of study medication.
Extubation time | Extubation
  Time for extubation of tracheal tube in minutes
Visual Analogue Scale VAS of Pain intensity | VAS (visual analogue scale) at 1, 2, 4, 8, 12 and 24 hours postoperatively.
  Pain scale measurement for postoperative assessment of pain consisting from 0 to 10 representing 0 as no pain and 10 as the most imaginable pain treating the patient if VAS > 3

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elsadany, MD, Principal Investigator — Anesthesia Department, Faculty of Medicine, Suez Canal University

IPD SHARING:
Plan to Share IPD: Undecided